CLINICAL TRIAL: NCT02254044
Title: An Open Phase I Dose Escalation Study of Bivatuzumab Mertansine Administered Intravenously Once Per Week for Three Weeks in Patients With Advanced Squamous Cell Carcinoma of the Head and Neck or Esophagus With Repeated Administration Courses in Patients With Clinical Benefit
Brief Title: Dose Escalation of Bivatuzumab Mertansine in Patients With Advanced Squamous Cell Carcinoma of the Head and Neck or Esophagus
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1191.4
Record Dates: First submitted 2014-09-30; First posted 2014-10-01 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Carcinoma, Squamous Cell
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — bivatuzumab mertansine

ARMS (1):
- bivatuzumab mertansine (Experimental): dose escalation
  Interventions: Drug: bivatuzumab mertansine

INTERVENTIONS:
Drug: bivatuzumab mertansine

SUMMARY:
maximum tolerated dose (MTD), safety, pharmacokinetics, efficacy of bivatuzumab mertansine

ELIGIBILITY:
Inclusion Criteria:

1. patients from 18 to 80 years of age (both inclusive)
2. patients with histologically confirmed squamous cell carcinoma of the head and neck or esophagus
3. patients with local and / or regional recurrent disease or distant metastases who are refractory to or not amenable to established treatments
4. evaluable tumour deposits
5. life expectancy of at least 3 months
6. Eastern Cooperative Oncology Group (ECOG) performance score ≤ 2
7. patients must have given written informed consent (which must be consistent with International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation)

Exclusion Criteria:

1. hypersensitivity to humanised or murine antibodies, immunoconjugates or the excipients of the trial drugs
2. known secondary malignancy requiring therapy
3. active infectious disease
4. brain metastases requiring therapy
5. neuropathy grade 2 or above
6. absolute neutrophil count less than 1,500/mm3
7. platelet count less than 100,000/mm3
8. bilirubin greater than 1.5 mg/dl (> 26 μmol/L, système internationale (SI) unit equivalent)
9. aspartate amino transferase (AST) and/or alanine amino transferase (ALT) greater than 3 times the upper limit of normal
10. serum creatinine greater than 1.5 mg/dl (> 132 μmol/L, SI unit equivalent)
11. concomitant non-oncological diseases which are considered relevant for the evaluation of the safety of the trial drug
12. chemo-, radio- or immunotherapy within the past four weeks prior to treatment with the trial drug or during the trial (except for present trial drug)
13. men and women who are sexually active and unwilling to use a medically acceptable method of contraception
14. pregnancy or lactation
15. treatment with other investigational drugs or participation in another clinical trial within the past four weeks before start of therapy or concomitantly with this trial (except for present trial drug)
16. patients unable to comply with the protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2003-10; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | up to 6 months

SECONDARY OUTCOMES:
Incidence of adverse events | up to 14 days after last drug administration
  graded according to common toxicity criteria (CTC)
Number of patients with clinically significant findings in laboratory examinations | up to 14 days after last drug administration
Number of patients with clinically significant findings in vital signs | up to 14 days after last drug administration
Number of patients with development of Human Anti-Human Antibody (HAHA) | up to 14 days after last drug administration
Area under the serum concentration time curve from time zero to time point 168 hours (AUC0-168) | up to 168 hours
Area under the serum concentration time curve from time zero to the time of the last quantifiable drug concentration (AUC0-tz) | up to 14 days after last drug administration
Area under the serum concentration time curve from time point zero to infinity (AUC0-∞) | up to 14 days after last drug administration
Maximum serum concentration (Cmax) | up to 14 days after last drug administration
Time to reach maximum serum concentration (tmax) | up to 14 days after last drug administration
Terminal elimination half-life (t1/2) | up to 14 days after last drug administration
Mean residence time (MRT) | up to 14 days after last drug administration
Total body clearance (CL) | up to 14 days after last drug administration
Volume of distribution at steady state (Vss) | up to 14 days after last drug administration
Volume of distribution during the terminal elimination phase (Vz) | up to 14 days after last drug administration
Trough concentration at steady state (Cpre,ss) | up to 7 days after drug administration
Minimum serum concentration during the dosing interval τ at steady state (Cmin,ss) | up to 7 days after drug administration
Linearity index (LI) | up to 14 days after last drug administration
Accumulation factor (RA) | up to 14 days after last drug administration
Tumor response | up to 14 days after last drug administration
  according to response evaluation criteria in solid tumours (RECIST)